CLINICAL TRIAL: NCT00507819
Title: The Sildenafil After Fontan Operation Study
Brief Title: Sildenafil After the Fontan Operation
Acronym: SAFO
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: The Mark H. and Blanche M. Harrington Foundation (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB 2007-4-5034
Record Dates: First submitted 2007-07-25; First posted 2007-07-27 (Estimated); Results first posted 2015-05-05 (Estimated); Last update posted 2015-05-05 (Estimated); Status verified 2015-05

CONDITIONS: Hypoplastic Left Heart Syndrome; Tricuspid Atresia
Keywords: Other Single Ventricle Anatomy; Hypoplastic Left Heart Syndrome; Tricuspid Atresia
MeSH Terms: conditions — Hypoplastic Left Heart Syndrome; Tricuspid Atresia | interventions — Sildenafil Citrate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sildenafil, then Placebo (Active Comparator): Sildenafil will be given at a dose of 20 mg three times-a-day for six weeks followed by a six week washout period followed by placebo for an additional six weeks.
  Interventions: Drug: Sildenafil; Drug: Placebo
- Placebo, then Sildenafil (Active Comparator): Placebo will be given for six weeks followed by a six week washout period followed by Sildenafil which will be given at a dose of 20 mg three times-a-day for six weeks
  Interventions: Drug: Sildenafil; Drug: Placebo

INTERVENTIONS:
Drug: Sildenafil — One 20 mg capsule of sildenafil will be taken by mouth three times-a-day.
  Other Names: Revatio; Viagra
Drug: Placebo — One placebo capsule will be taken by mouth three times-a-day.

SUMMARY:
In this study, the investigators will evaluate the effect of sildenafil on exercise tolerance in patients with a single cardiac ventricle who have undergone the Fontan operation. The investigators will also evaluate echocardiographic measures of ventricular function and measure quality of life changes using two validated quality of life measures. The hypothesis is that sildenafil will result in increased exercise tolerance in patients who have had the Fontan operation as compared to placebo.

DETAILED DESCRIPTION:
The Fontan physiology is the end result of staged reconstruction of the heart and the major blood vessels in patients who have a single ventricle. After completion of the reconstruction, the great veins which usually bring blood back to the heart are connected directly to the pulmonary arteries, allowing blood from the body to bypass the heart and flow directly into the lungs. In this system, blood flow through the lungs is passive (not pumped) and the efficiency of flow through the cardiovascular system is related to the resistance to blood flow in the vessels of the lungs.

There are two potential problems that arise in this scenario, as a result of the resistance to blood flow in the vessels of the lungs. First, the amount of blood flow returning to the heart from the lungs may not be sufficient to allow the heart to function at maximum efficiency, compromising the heart's ability to keep up with the demands of the body. Second, if the resistance to blood flow in the lungs is high, pressure may be transmitted back into the great veins themselves and secondarily into the organs of the body causing mild, or sometimes significant, organ dysfunction. Not all patients with the Fontan physiology develop these problems, but we know that even in patients without obvious problems, the ability to keep up with an increased metabolic demand, as during exercise, in compromised.

Improving the efficiency of blood flow through the lungs should improve the return of blood to the heart and thereby diminish the pressure transmitted back to the vessels which passively deliver blood to the lungs. We believe that this change may manifest as diminished symptoms in those patients with known difficulties, or may allow for an increased ability to walk, run, or participate in sports in those without any overt symptoms. Most importantly, we speculate that improved efficiency of flow through the lungs, and the resulting improved cardiac output (blood flow through the body) will make patients more energetic and will make them feel better.

Sildenafil is an oral medication that has been used to treat patients with pulmonary hypertension, a disease in which there is abnormally elevated pressure in the vessels of the lung. In this disease, the resistance in the lungs is abnormally high, severely limiting the ability of the heart to keep up with the demands of the body. Sildenafil lowers the resistance in the vessels of the lungs and has been shown to improve exercise performance in patients with this disease. We believe that Sildenafil may have a similar benefit for our patients after Fontan operation in whom cardiac output is also limited by resistance of the blood vessels in the lungs.

In our study, we will compare the exercise capacity, echocardiographic measures of cardiac function, and the overall quality of life in patients with the Fontan before and after a six-week period of sildenafil administration. As a control, the same group of patients will take a placebo for a six-week period, also with before and after testing. We hypothesize that oral sildenafil will result in significant improvements in exercise capacity, energy levels, and echocardiographic measures of cardiac function and output in our study participants. We are hopeful that the findings of this investigation will directly help children and young adults with Fontan physiology.

ELIGIBILITY:
Inclusion Criteria:

* 8 years of age or older
* All participants must have had Fontan completion

Exclusion Criteria:

* Height less than 132 cm
* Unable to participate in exercise testing due to medical restrictions or physical limitations
* Fontan baffle obstruction or single lung physiology
* Coarctation of the aorta or neo-aorta (BP gradient > 20 mmHg)
* Severe ventricular dysfunction assessed qualitatively by echocardiography
* Severe atrioventricular valvar regurgitation assessed qualitatively by echocardiography
* Presence of electronic pacemaker
* History of treatment with sildenafil in the six weeks prior to enrollment in study
* Patients with severe renal impairment
* Patients with severe hepatic impairment
* Patients taking medications that inhibit or induce Cytochrome P450 3A4 (CYP3A4) (including grapefruit juice and St. John's Wort)
* Patients taking alpha-blockers and nitrates
* Parents/guardians or subjects who, in the opinion of the investigator, may be non-compliant with study schedules or procedures

Ages: 8 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 28 (Actual)
Dates: Start 2007-12; Primary Completion 2009-04 (Actual); Study Completion 2009-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jack Rychik, MD, Principal Investigator — Children's Hospital of Philadelphia

REFERENCES:
- [Derived] Goldberg DJ, French B, McBride MG, Marino BS, Mirarchi N, Hanna BD, Wernovsky G, Paridon SM, Rychik J. Impact of oral sildenafil on exercise performance in children and young adults after the fontan operation: a randomized, double-blind, placebo-controlled, crossover trial. Circulation. 2011 Mar 22;123(11):1185-93. doi: 10.1161/CIRCULATIONAHA.110.981746. Epub 2011 Mar 7. PMID 21382896

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Of 125 eligible subjects contacted by the study team, 28 (22%) participated in the study.
Groups:
- Placebo, Then Sildenafil: Placebo six weeks followed by a six week washout period followed by Sildenafil which will be given at a dose of 20 mg three times-a-day for six weeks
Period: First Intervention (6 Weeks)
Arm/Group | Sildenafil, Then Placebo | Placebo, Then Sildenafil
Started | 14 | 14
Completed | 14 | 14
Not Completed | 0 | 0
Period: Washout (6 Weeks)
Arm/Group | Sildenafil, Then Placebo | Placebo, Then Sildenafil
Started | 14 | 14
Completed | 13 | 14
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0
Period: Second Intervention (6 Weeks)
Arm/Group | Sildenafil, Then Placebo | Placebo, Then Sildenafil
Started | 13 | 14
Completed | 13 | 14
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: All subjects who consented to participate and were randomized, completed at least the first six-week study period.
Groups:
- Study Population: Subjects who were randomized to receive either Sildenafil 20mg three times a day by mouth or Placebo three times a day by mouth.
Arm/Group | Study Population
Number analyzed (Participants) | 28
Age, Continuous [Mean (Standard Deviation); unit: Years] | 14.9 (5.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 18

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Mean Oxygen Consumption (mL/kg/Min) at 6 Weeks
Description: Oxygen consumption measurements were taken at peak exercise. Subjects were exercised to maximal volition with an electronically braked cycle ergometer. The protocol consisted of 3 minutes of pedaling in an unloaded state followed by a ramp increase in work rate (watts) to maximal exercise. Metabolic and ventilatory data were obtained throughout the exercise study and for the first 2 minutes of recovery on a breath-by-breath basis with a metabolic cart.
Time Frame: Baseline and 6 Weeks
Measure: Mean (Standard Deviation); unit: mL/kg/min
Groups:
- Sildenafil: Sildenafil was given by mouth at a dose of 20 mg three times a day for six weeks
- Placebo: Placebo was given by mouth three times a day for six weeks
Arm/Group | Sildenafil | Placebo
Number analyzed (Participants) | 28 | 27
mL/kg/min
  Oxygen Consumption at Baseline (mL/kg/min) | 30.5 (6.9) | 30.5 (6.9)
  Oxygen Consumption at 6 Weeks (mL/kg/min) | 31.3 (7.1) | 31.3 (7.5)
Statistical Analysis 1: Comparison: Sildenafil vs Placebo; Test type: Superiority or Other; p = 0.73, Regression, Linear

2. Secondary Outcome: Change From Baseline in Mean Heart Rate (Bpm) at 6 Weeks
Description: Heart rate was measured at peak exercise. Subjects were exercised to maximal volition with an electronically braked cycle ergometer. The protocol consisted of 3 minutes of pedaling in an unloaded state followed by a ramp increase in work rate (watts) to maximal exercise. Metabolic and ventilatory data were obtained throughout the exercise study and for the first 2 minutes of recovery on a breath-by-breath basis with a metabolic cart.
Time Frame: Baseline and 6 Weeks
Measure: Mean (Standard Deviation); unit: bpm
Arm/Group | Sildenafil | Placebo
Number analyzed (Participants) | 28 | 27
bpm
  Heart rate at Baseline (bpm) | 163 (20) | 163 (15)
  Heart rate at 6 Weeks (bpm) | 163 (14) | 163 (15)
Statistical Analysis 1: Comparison: Sildenafil vs Placebo; Test type: Superiority or Other; p = 0.37, Regression, Linear

3. Secondary Outcome: Change From Baseline in Mean Respiratory Rate (Breaths/Min) at 6 Weeks
Description: Respiratory rate was measured at peak exercise. Subjects were exercised to maximal volition with an electronically braked cycle ergometer. The protocol consisted of 3 minutes of pedaling in an unloaded state followed by a ramp increase in work rate (watts) to maximal exercise. Metabolic and ventilatory data were obtained throughout the exercise study and for the first 2 minutes of recovery on a breath-by-breath basis with a metabolic cart.
Time Frame: Baseline and 6 Weeks
Measure: Mean (Standard Deviation); unit: breaths/min
Arm/Group | Sildenafil | Placebo
Number analyzed (Participants) | 28 | 27
breaths/min
  Mean Respiratory rate at Baseline (breaths/min) | 53.7 (8.9) | 53.0 (7.5)
  Mean Respiratory rate at 6 Weeks (breaths/min) | 51.0 (9.4) | 53.0 (8.3)
Statistical Analysis 1: Comparison: Sildenafil vs Placebo; Test type: Superiority or Other; p = 0.05, Regression, Linear

4. Secondary Outcome: Change From Baseline in Mean Minute Ventilation (L/Min) at 6 Weeks
Description: Minute ventilation measurements were taken at peak exercise. Subjects were exercised to maximal volition with an electronically braked cycle ergometer. The protocol consisted of 3 minutes of pedaling in an unloaded state followed by a ramp increase in work rate (watts) to maximal exercise. Metabolic and ventilatory data were obtained throughout the exercise study and for the first 2 minutes of recovery on a breath-by-breath basis with a metabolic cart.
Time Frame: Baseline and 6 Weeks
Measure: Mean (Standard Deviation); unit: L/min
Arm/Group | Sildenafil | Placebo
Number analyzed (Participants) | 28 | 27
L/min
  Minute Ventilation at Baseline (L/min) | 68.8 (25) | 68.1 (27)
  Minute Ventilation at 6 Weeks (L/min) | 67.2 (23) | 68.8 (26)
Statistical Analysis 1: Comparison: Sildenafil vs Placebo; Test type: Superiority or Other; p = 0.04, Regression, Linear

ADVERSE EVENTS:
Time Frame: 6 weeks for each intervention.
Description: Adverse event summary information includes all subjects who received at least one dose of study medication/placebo.
Arm/Group | Sildenafil | Placebo
Serious Adverse Events (participants affected / at risk) | 1/28 | 0/27
Other Adverse Events (participants affected / at risk) | 11/28 | 10/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sildenafil (N=28) | Placebo (N=27)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) — Constipation-related abdominal pain
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sildenafil (N=28) | Placebo (N=27)
Headache (General disorders) | 9 (9) | 5 (5) — Headache
Flushing (Vascular disorders) | 5 (5) | 0 (0) — Non-painful facial flushing
Dizziness (General disorders) | 2 (2) | 2 (2) — Dizziness
Nausea / vomiting (Gastrointestinal disorders) | 2 (2) | 0 (0) — Nausea / vomiting
Kidney Stone (Renal and urinary disorders) | 1 (1) | 0 (0)
Photosensitivity (Eye disorders) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hypotension (Cardiac disorders) | 0 (0) | 1 (1)
Muscle Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Tremulous (General disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Characteristics of screened but not enrolled subjects was not evaluated, so enrolled subjects may not be a representative sample from the group at large. Safety of Sildenafil over a prolonged (>6week) period of continuous use was not evaluated.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No